CLINICAL TRIAL: NCT06447376
Title: Pilot Safety-feasibility Study of Cytokine Release Syndrome Prophylaxis and Treatment With Siltuximab Prior to Epcoritamab
Brief Title: Study of Cytokine Release Syndrome Prophylaxis and Treatment With Siltuximab Prior to Epcoritamab
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taylor Brooks (Other)
Collaborators: Genmab (Industry); AbbVie (Industry); RECORDATI GROUP (Industry)
Responsible Party: Sponsor-Investigator, Taylor Brooks, IND Holder, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1424
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Non-Hodgkin Lymphoma; Cytokine Release Syndrome
Keywords: Siltuximab; Epcoritamab; Prophylactic siltuximab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Cytokine Release Syndrome | interventions — siltuximab

STUDY DESIGN:
Intervention Model Description: Single cohort study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prophylactic siltuximab + epcoritamab (Experimental): Siltuximab Administration:
  • Participants will receive a single dose of prophylactic siltuximab, 11mg/kg, started 1 hour prior (+/- 60 minutes) to the infusion of epcoritamab. There is no planned dose escalation of siltuximab and epcoritamab dosing will be done following the standard planned ramp-up over the course of the first 3 weeks
  Epcoritamab Infusion:
  • The treatment regimen of epcoritamab is done in 28-day cycles. Epcoritamab is to be administered by subcutaneous injection. Participants can be treated for up to 24 cycles. Participants who achieve complete remission at the time of their disease response assessment after 12 cycles may be considered for early discontinuation of treatment.
  Interventions: Drug: Siltuximab; Drug: Epcoritamab

INTERVENTIONS:
Drug: Siltuximab — Single dose of prophylactic siltuximab, 11mg/kg, started 1 hour prior (+/- 60 minutes) to the infusion of epcoritamab.
Drug: Epcoritamab — Epcoritamab dosing for Diffuse Large B-cell Lymphoma Participants:
  * Cycle 1, Day 1 = 0.16mg
  * Cycle 1, Day 8 = 0.8mg
  * Cycle 1, Day 15 = 48mg
  * Cycle 1, Day 22 = 48mg
  * Cycles 2 & 3, Day 1 = 48mg
  * Cycles 2 & 3, Day 8 = 48mg
  * Cycles 2 & 3, Day 15 = 48mg
  * Cycles 2 & 3, Day 22 = 48mg
  * Cycles 4-9, Day 1 = 48mg
  * Cycles 4-9, Day 15 = 48mg
  * Cycle 10+ , Day 1 = 48mg
  Epcoritamab dosing for Follicular Lymphoma Participants:
  * Cycle 1, Day 1 = 0.16mg
  * Cycle 1, Day 8 = 0.8mg
  * Cycle 1, Day 15 = 3mg
  * Cycle 1, Day 22 = 48mg
  * Cycle 2 & 3, Day 1 = 48mg
  * Cycle 2 & 3, Day 8 = 48mg
  * Cycle 2 & 3, Day 15 = 48mg
  * Cycle 2 & 3, Day 22 = 48mg
  * Cycle 4-9, Day 1 = 48mg
  * Cycle 4-9, Day 15 = 48mg
  * Cycle 10+ , Day 1 = 48mg

SUMMARY:
The goal of this clinical trial is to is to determine the safety, feasibility and efficacy of siltuximab prophylaxis of cytokine release syndrome and neurotoxicity occurring after epcoritamab subcutaneous administration for participants with large b-cell lymphoma (DLBCL) or follicular lymphoma (FL).

Participants will receive siltuximab, prior to the injection of epcoritamab. Epcoritamab is administered in 28 day cycles for one year. After this injection, the physician will continue to watch participants for side effects and follow the condition for a minimum of 60 days.

DETAILED DESCRIPTION:
Siltuximab is a monoclonal antibody that blocks interleukin-6 (IL-6) from binding to its receptor, preventing it from acting. IL-6 is a cytokine, a type of protein that is a cause of inflammatory reactions. Decreasing levels of IL-6 has been shown to reduce symptoms of cytokine release syndrome (CRS), a potential side effect of epcoritamab. Addition of siltuximab to the medications given before epcoritamab, may prevent, or reduce the severity, of CRS. Siltuximab is experimental because it is not approved by the Food and Drug Administration for treatment or prevention of CRS. Epcoritamab is a so-called bispecific antibody, which is a molecule that can bind simultaneously to two different receptors. Epcoritamab binds to a receptor called CD3 with one part of the antibody and to a receptor called CD20 with another part of the antibody. CD20 is expressed on the normal, healthy B cells but also on the cancerous lymphoma cells of B cell origin. CD3 is expressed on T cells, which are important cells of the immune system and help the body fight cancers, infections, etc. By simultaneous binding to CD3 and CD20, Epcoritamab brings T cells and B cells close together and activates the T cells to kill the B cells, including the cancerous ones.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and older
* Diagnosis of non-Hodgkin lymphoma.

  * DLBCL (including high grade B cell lymphoma and follicular lymphoma grade 3B and transformed follicular lymphoma) treated with at least 2 lines of systemic antineoplastic therapies, including at least 1 anti-CD20 monoclonal antibody - containing therapy
  * FL grade 1-3A previously treated with at least 2 lines of systemic antineoplastic therapy, including at least 1 anti-CD20 monoclonal antibody - containing therapy.
* At least 1 risk factor for cytokine release syndrome, including:

  * Age ≥ 65 years,
  * Elevated lactate dehydrogenase,
  * White blood cell count pre-anti-CD20 treatment > 4.5x109 cells/L,
  * Ann Arbor Stage III/IV,
  * Sum of the product of the perpendicular diameters at study entry ≥3000mm2,
  * Cardiac comorbidity, including prior coronary disease, heart failure and other conditions that in the opinion of the investigator would increase the risk of heightened toxicity from CRS
  * Bone marrow infiltration,
  * Circulating lymphoma cells in peripheral blood
* Adequate bone marrow function including:

  * Hemoglobin ≥ 8g/dL (unless bone marrow involvement by lymphoma) (transfusion allowed for symptomatic participants),
  * Absolute neutrophil count cell count ≥1000 / μL, with or without growth factor support
  * Platelet counts ≥ 75,000 / μL (unless bone marrow involvement by lymphoma, in which case platelet counts ≥ 50,000 / µL are required)
* ECOG performance status 0 - 2
* Creatinine clearance ≥ 30 mL/min
* Adequate hepatic function:

  * AST and/or ALT up to 3 times upper limit of normal (unless elevation is secondary to disease involvement of the liver, in which case up to 5 times upper limit is permitted after discussion with the principal investigator).
  * Total bilirubin up to 1.5 times upper limit of normal (unless elevation is secondary to Gilbert syndrome or of non - hepatic origin).
* Subjects (or legal guardians) must have the ability to understand and the willingness to sign a written informed consent document.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (< 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period. Men must refrain from donating sperm during this same period. With pregnant female partners, men must remain abstinent or use a condom during the treatment period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Primary mediastinal B cell lymphoma
* Active central nervous system or meningeal involvement by lymphoma
* History of severe allergic or anaphylactic reactions to anti-CD20 monoclonal antibody therapy
* Active bacterial, viral, fungal, mycobacterial, parasitic or other infection requiring systemic therapy within 2 weeks prior to first dose of study drug. This includes participants with COVID-19 infection
* History of active chronic infection by hepatitis B or C or Cytomegalovirus (CMV) requiring treatment or prophylaxis. Resolved infections (either by treatment or immune response) are not exclusion criterion.
* Active malignancy, other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast). History of prior malignancy is not excluded.
* HIV seropositivity.
* Subjects with uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because siltuximab therapy may be associated with the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative serum pregnancy test. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with siltuximab, breastfeeding should be continued and not restarted for 3 months after the last dose of siltuximab. These potential risks may also apply to other agents used in this study.
* Participants with history of clinically relevant and active CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of all-grade cytokine release syndrome | Up to 28 days after beginning treatment
  The primary objective is to evaluate the feasibility and efficacy of prophylactic administration of siltuximab prior to infusion of the first dose of epcoritamab with the purpose of preventing all-grade CRS, as measured by incidence of all-grade cytokine release syndrome.

SECONDARY OUTCOMES:
Incidence of grade ≥ 2 cytokine release syndrome | Up to 28 days after beginning treatment
  A secondary objective is to determine the incidence of grade ≥ 2 CRS after siltuximab prophylaxis
Incidence of all grade and grade ≥ 2 ICANS after siltuximab prophylaxis | Up to 28 days beginning treatment
  A secondary objective is to determine the incidence of all grade and grade ≥ 2 ICANS after siltuximab prophylaxis
Incidence of adverse events during Cycle 1 (Day 1 - 28) | Up to 28 days after beginning treatment
  A secondary objective is to describe the adverse events after siltuximab prophylaxis.
Best overall and complete response rates | Up to 456 days after beginning treatment
  A secondary objective is to describe the disease response rates (overall and complete response rates) to epcoritamab in participants treated with prophylactic siltuximab, based on Lugano response criteria for malignant lymphomas, which can include complete response (CR), partial response (PR), stable disease (SD), progression (PD) and relapse.
Incidence of hospitalizations secondary to all causes | Up to 456 days after beginning treatment
  A secondary objective is to describe the rates of hospitalization for all causes and for cytokine release syndrome
Incidence of hospitalizations secondary to cytokine release syndrome or neurologic complications | Up to 456 days after beginning treatment
  A secondary objective is to describe the rates of hospitalization for for cytokine release syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Taylor Brooks, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared with the FDA and Recordati and Genmab who are the suppliers of the investigational products any participant data shared will be deidentified.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available during the course of the trial and indefinitely thereafter.
Access Criteria: Data will be available for the FDA otherwise a confidentiality agreement will need to be in place